CLINICAL TRIAL: NCT01923623
Title: The Effect of Combined Popliteal and Saphenous Block in Addition to General Anesthesia in Surgical Fixation of Ankle Fractures: a Prospective Randomized Study
Brief Title: The Effect of Nerve Blockades in Addition to General Anesthesia in Surgical Fixation of Ankle Fractures.
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Study was redesigned and taken over by a ph.D-student
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Heidi Kruse, Pregraduat research assistent, Herlev Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: Huggi123
Record Dates: First submitted 2013-08-13; First posted 2013-08-15 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-04

CONDITIONS: Ankle Fracture in Need of Surgical Fixation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Block (Experimental): Popliteal and saphenous Block with Ropivacaine
  Interventions: Drug: Ropivacaine block
- NaCl (Placebo Comparator)
  Interventions: Drug: Ropivacaine block

INTERVENTIONS:
Drug: Ropivacaine block

SUMMARY:
This clinical, randomized, and controlled study will provide valuable scientific evidence regarding the effect of adding peripheral nerve blockades to general anaesthesia during ankle surgery. In particular, the investigators want to determine if the need for postoperative opioids will be reduced and whether this will lead to shorter admission to recovery room and fewer instances of side effects such as postoperative nausea and vomiting. In addition, the investigators will determine whether the functional outcome is improved i.e. faster and more successful rehabilitation. This would have profound benefits not only to the individual patient but also to society by reducing expenses during admission, the cost of sick leave etc.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Patients in need of anaesthesia for operative fixation of ankle fractures.
* American Society of Anesthesiologists (ASA) score 1-3.
* BMI > 18 og < 35.
* Oral and written consent

Exclusion Criteria:

* Weight < 50kg
* Allergy towards drugs used in the study
* Patients for re-operation
* Other fracture at the same time
* Pregnancy
* Daily use of opioids within two weeks before operation
* Infection near the application site
* Patients in need of dialysis
* Patients with neuropathy in lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-07-01 (Actual); Primary Completion 2013-07-01 (Actual); Study Completion 2013-07-31 (Actual)

PRIMARY OUTCOMES:
Use of Morphine | 24 hours

SECONDARY OUTCOMES:
Functional rehabilitation outcome | 10-14 weeks
  American Orthopaedic Foot and Ankle Society (AOFAS) score

CONTACTS AND LOCATIONS:
Overall Officials: Rune Sort, M.D., Principal Investigator — Herlev Hospital; Ann M. Møller, Dr.med., Study Director — Herlev Hospital